CLINICAL TRIAL: NCT04195269
Title: Osteoarthritis of the Knee Pain Study Using CBD and THC in Rapidly Dissolvable Sublingual Tablet
Brief Title: Osteoarthritis of the Knee Pain Study Using a CBD and THC Sublingual Tablet
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Pure Green (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: PG-OA-1010-19-004
Record Dates: First submitted 2019-12-09; First posted 2019-12-11 (Actual); Last update posted 2020-04-14 (Actual); Status verified 2020-04

CONDITIONS: Osteoarthritis, Knee; Pain
Keywords: CBD; THC; Cannabidiol; Tetrahydrocannabinol; Osteoarthritis; Knee; Pain
MeSH Terms: conditions — Osteoarthritis, Knee; Pain; Osteoarthritis

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Pure Green Sublingual Tablet - Daily (Experimental): Subjects will take 2 tablets daily, one in the morning and one in the evening, and are able to take up to 2 additional tablets per day as needed for pain.
  Interventions: Drug: Test Article

INTERVENTIONS:
Drug: Test Article — 10 mg CBD, 10 mg of THC, and a proprietary blend of terpenes.

SUMMARY:
This study is a prospective Phase 2, drug controlled, open-label study to evaluate the safety and efficacy of Pure Green sublingual tablets for the treatment of pain associated with osteoarthritis of the knee.

ELIGIBILITY:
Inclusion Criteria:

1. Subject is at least 21 years of age;
2. Subject has a diagnosis of a pain related to osteoarthritis of the knee as determined by the subject's primary care physician or related health care provider.
3. Subject has a mean pain scale score of ≥ 4 recorded in the 7 days prior to enrollment.
4. If female, the subject is postmenopausal (> 1 year), surgically sterile (> 3 months), had a hysterectomy, or is currently using 2 effective forms of birth control.
5. Subject has not taken marijuana (cannabis) in any form, chemicals or extracts or foods or beverages or topical creams, lotions, gels, patches containing marijuana (cannabinoids, or and cannabis derivatives) including synthetic marijuana and/or CBD for at least 14 days prior to this study, and promises to not take marijuana (cannabis) in any form, chemicals or extracts or foods or beverages or topical creams, lotions, gels, patches containing marijuana (cannabinoids, or and cannabis derivatives) including synthetic marijuana and/or CBD while participating in this study.
6. Subject has not taken any pain medication, including NSAIDs, for at least 2 days before taking the first dose of study drug.
7. Subject is willing to provide his/her written informed consent to participate in the study as stated in the informed consent document.
8. Subject is willing to use an electronic diary to enter a pain scale score up to four times a day for 28 days.

Exclusion Criteria

1. Subject is pregnant or lactating;
2. Subject has an allergy to cannabis, the Cannabaceae plant family (e.g., hemp, hops), palmitoylethanolamide, or terpenes;
3. Subject has a known allergy to active or inert ingredients of PG-OA-10:10-2020-B tablets;
4. Subject is taking a concomitant medication or treatment that would complicate use or interpretation of the study drug's effects (examples include: Cannabis or any cannabinoid products; Any drug or herbal product that influences the endocannabinoid system (ECS));
5. Subject is taking marijuana (cannabis) in any form, chemicals or extracts or foods or beverages or topical creams, lotions, gels, patches containing marijuana (cannabinoids, or and cannabis derivatives) including synthetic marijuana and/or CBD for at least 14 days prior to this study, and does not promise that they will not take marijuana (cannabis) in any form, chemicals or extracts or foods or beverages or topical creams, lotions, gels, patches containing marijuana (cannabinoids, or and cannabis derivatives) including synthetic marijuana and/or CBD while participating in this study;
6. Subject is currently being treated with antibiotics for sinus, throat, or lung infections;
7. Subject has shortness of breath associated with allergies;
8. Subject has uncontrolled asthma;
9. Subject has a fever and/or productive cough;
10. Subject has unstable angina, uncontrolled hypertension;
11. Subject currently or has a history of congestive heart failure;
12. Subject has any other unstable medical condition;
13. Subject has a personal or family history of schizophrenia;
14. Subject has a personal history or currently has suicidal ideation or attempted suicide;
15. Subject has a major neurological disorder, such as dementia, Parkinson's disease, cognitive impairment, epilepsy, history of traumatic brain injury/head injury, and seizures.
16. Subject has taken pain medicine of any kind throughout the screening period, or has taken acetaminophen within 2 days of taking the first dose of study drug.
17. Subject has an allergy to, or has an intolerance to, acetaminophen.
18. Subject is currently taking any form of opioids.
19. Subject has a history of alcohol or substance abuse
20. Subject has clinically significant illness, including cardiovascular disorders.
21. Subject has any condition in which the investigator believes will confound the data of the study or could put the subject at risk of harm.
22. Subject does not have access to a smart phone or does not know how to use a smart phone application.

Min Age: 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2020-04-20 (Estimated); Primary Completion 2020-06-30 (Estimated); Study Completion 2020-07-15 (Estimated)

PRIMARY OUTCOMES:
Impact of Pure Green sublingual tablets on pain due to osteoarthritis of the knee using a daily self-reported pain scale score. | 30 days
  To evaluate the safety and efficacy of Pure Green sublingual tablets for the treatment of pain due to osteoarthritis of the knee by having patients evaluate their daily pain scale score reported as 0-10 where 0 is no pain and 10 is the worst pain possible as self-reported with every dose taken by the patient in the smart phone app. The objective is to reduce the patients average daily pain scale score to less than 4.

SECONDARY OUTCOMES:
Impact of Pure Green sublingual tablets on general health and well-being of Osteoarthritis of the knee patients. | 30 Days
  To evaluate the impact of Pure Green sublingual tablets on the general health and well-being of osteoarthritis of the knee patiens. The objective is to examine quality of life metrics: overall quality of life and general health, physical health, and knee pain as measured on a 1-5 scale before and after the study
Impact of Pure Green sublingual tablets on sleep improvement of patients with osteoarthritis of the knee. | 30 Days
  The Pittsburgh Sleep Quality Index will be used to compare pre and post Pure Green sublingual tablet study on sleep changes. Patients will be asked questions before beginning of the study and after completion.
Impact of Pure Green sublingual tablets on anxiety of patients with osteoarthritis if the knee | 30 Days
  The Hamilton Anxiety rating scale questionnaire will be administered before the study begins and after completion to examine the impact of Pure Green sublingual tablets on anxiety in patients with osteoarthritis of the knee. The scale of 0-4 will be used where 0 is no anxiety present and 4 is very severe anxiety.
Impact on the use of sublingual tablets as the route of administration. | 30 Days
  To explore the impact of sublingual administration on patient compliance by evaluating the number of tablets taken per day as entered by the patients into the smart phone app.

CONTACTS AND LOCATIONS:
Overall Officials: Debra Kimless, M.D., Principal Investigator — Chief Medical Officer
Locations (1):
- Pure Green, LLC, West Bloomfield, Michigan, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Brown JP, Boulay LJ. Clinical experience with duloxetine in the management of chronic musculoskeletal pain. A focus on osteoarthritis of the knee. Ther Adv Musculoskelet Dis. 2013 Dec;5(6):291-304. doi: 10.1177/1759720X13508508. PMID 24294303
- [Background] Blake DR, Robson P, Ho M, Jubb RW, McCabe CS. Preliminary assessment of the efficacy, tolerability and safety of a cannabis-based medicine (Sativex) in the treatment of pain caused by rheumatoid arthritis. Rheumatology (Oxford). 2006 Jan;45(1):50-2. doi: 10.1093/rheumatology/kei183. Epub 2005 Nov 9. PMID 16282192
- [Background] Australian Public Assessment Report for Nabiximols
- [Background] O'Brien M, McDougall JJ. Cannabis and joints: scientific evidence for the alleviation of osteoarthritis pain by cannabinoids. Curr Opin Pharmacol. 2018 Jun;40:104-109. doi: 10.1016/j.coph.2018.03.012. Epub 2018 Apr 7. PMID 29635215
- [Background] Huggins JP, Smart TS, Langman S, Taylor L, Young T. An efficient randomised, placebo-controlled clinical trial with the irreversible fatty acid amide hydrolase-1 inhibitor PF-04457845, which modulates endocannabinoids but fails to induce effective analgesia in patients with pain due to osteoarthritis of the knee. Pain. 2012 Sep;153(9):1837-1846. doi: 10.1016/j.pain.2012.04.020. Epub 2012 Jun 21. PMID 22727500
- [Background] Fukuda S, Kohsaka H, Takayasu A, Yokoyama W, Miyabe C, Miyabe Y, Harigai M, Miyasaka N, Nanki T. Cannabinoid receptor 2 as a potential therapeutic target in rheumatoid arthritis. BMC Musculoskelet Disord. 2014 Aug 12;15:275. doi: 10.1186/1471-2474-15-275. PMID 25115332
- [Background] Krustev E, Reid A, McDougall JJ. Tapping into the endocannabinoid system to ameliorate acute inflammatory flares and associated pain in mouse knee joints. Arthritis Res Ther. 2014 Sep 27;16(5):437. doi: 10.1186/s13075-014-0437-9. PMID 25260980
- [Background] Smith FL, Fujimori K, Lowe J, Welch SP. Characterization of delta9-tetrahydrocannabinol and anandamide antinociception in nonarthritic and arthritic rats. Pharmacol Biochem Behav. 1998 May;60(1):183-91. doi: 10.1016/s0091-3057(97)00583-2. PMID 9610941
- [Background] Schuelert N, McDougall JJ. Cannabinoid-mediated antinociception is enhanced in rat osteoarthritic knees. Arthritis Rheum. 2008 Jan;58(1):145-53. doi: 10.1002/art.23156. PMID 18163511
- [Background] Schuelert N, Johnson MP, Oskins JL, Jassal K, Chambers MG, McDougall JJ. Local application of the endocannabinoid hydrolysis inhibitor URB597 reduces nociception in spontaneous and chemically induced models of osteoarthritis. Pain. 2011 May;152(5):975-981. doi: 10.1016/j.pain.2010.11.025. Epub 2010 Dec 24. PMID 21185649
- [Background] Richardson D, Pearson RG, Kurian N, Latif ML, Garle MJ, Barrett DA, Kendall DA, Scammell BE, Reeve AJ, Chapman V. Characterisation of the cannabinoid receptor system in synovial tissue and fluid in patients with osteoarthritis and rheumatoid arthritis. Arthritis Res Ther. 2008;10(2):R43. doi: 10.1186/ar2401. Epub 2008 Apr 16. PMID 18416822